CLINICAL TRIAL: NCT05487456
Title: A Randomized, Controlled, Open-label, 4-arm Parallel Group Study to Demonstrate Reductions in Exposure to Selected Harmful and Potentially Harmful Constituents (HPHC) in Healthy Smokers Switching to 2 Variants of P4M3 Gen 2.0, an Electronic Nicotine Delivery System (ENDS), Compared to Continuing Smoking Cigarettes, or Abstaining From Smoking, for 5 Days in a Confinement Setting
Brief Title: Reduced HPHC Exposure in Cigarette Smokers Switching to P4M3 Gen. 2.0 Compared to Continuing Smoking, or Smoking Abstinence
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Philip Morris Products S.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: P4-REXC-06
Record Dates: First submitted 2022-07-25; First posted 2022-08-04 (Actual); Results first posted 2024-03-13 (Actual); Last update posted 2024-03-13 (Actual); Status verified 2023-06

CONDITIONS: Nicotine; Vaping; Nicotine Vaping
Keywords: Nicotine; Smoking; Cigarette; E-Cigarette; Electronic Nicotine Delivery System; Vaping
MeSH Terms: conditions — Vaping; Smoking | interventions — Nicotine; Tobacco Products

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- P4M3 CA35 (Active Comparator): Ad libitum use of P4M3 using CA35 Cartridges
  Interventions: Other: P4M3 CA35
- P4M3 CM35 (Active Comparator): Ad libitum use of P4M3 using CM35 Cartridges
  Interventions: Other: P4M3 CM35
- Cigarette (Active Comparator): Ad libitum use of subject's own preferred CIG brand
  Interventions: Other: CIG
- Smoking Abstinence (Active Comparator): Smoking abstinence
  Interventions: Other: Smoking Abstinence

INTERVENTIONS:
Other: P4M3 CA35 — Ad libitum use of P4M3 with CA35 cartridges
  Other Names: P4M3 "Classic Auburn" 3.5% nicotine (CA35)
  Arms: P4M3 CA35
Other: P4M3 CM35 — Ad libitum use of P4M3 with CM35 cartridges
  Other Names: P4M3 "Classic Menthol" 3.5% nicotine (CM35)
  Arms: P4M3 CM35
Other: CIG — Ad libitum use of subject's own preferred brand of cigarettes
  Other Names: Cigarette
  Arms: Cigarette
Other: Smoking Abstinence — Abstention from cigarette smoking
  Arms: Smoking Abstinence

SUMMARY:
To demonstrate the reduction of Biomarkers of Exposure (BoExp) to selected harmful and potentially harmful constituents (HPHC) in smokers switching from cigarette (CIG) to P4M3, an Electronic Nicotine Delivery System (ENDS), compared to continuing cigarette smoking for 5 days.

DETAILED DESCRIPTION:
Reduced HPHC Exposure in Cigarette Smokers Switching to P4M3 Generation 2.0 Compared to Continuing Smoking, or Smoking Abstinence

* Who carried out the research? This research was sponsored and funded by Philip Morris Products S.A.
* What public involvement there was in the study? Sixty-eight healthy, currently smoking, adults participated in this study.
* Where and when the study took place? The study was conducted at a clinical trial facility managed by a contract research organization in Belfast, Northern Ireland, from July 15th to August 31st 2022.
* Why was the research needed? The research was needed to understand the reductions in exposure to selected harmful and potentially harmful constituents of cigarette smoke in healthy smokers, who switched exclusively to an electronic nicotine delivery system for five days.
* What were the main questions studied? The study measured the reductions in exposure to selected harmful and potentially harmful constituents of cigarette smoke in healthy smokers switching exclusively to two flavour variants (CA35 and CM35) of P4M3, an Electronic Nicotine Delivery System, compared to continued smoking of cigarettes or abstaining from smoking.
* Who participated in the study? Sixty-eight healthy, male or female, adults aged between 21 and 65 years participated in this study. All participants were currently smoking. The participants did not plan to quit using tobacco and/or nicotine products within the next 3 months and had smoked continuously for at least the last 3 years prior to joining the study. Each participant was given full and adequate oral and written information about the nature, purpose, possible risks, and benefits of the study. All participants received information on the risks of smoking, smoking cessation advice and a briefing on the P4M3 Electronic Nicotine Delivery System, for example, that its use is not risk-free. Once each participant had received all the necessary information, and if they agreed to participate, this was documented in an Informed Consent Form with the date, time and signature of both the participant and the study doctor. Participants were informed that they were free to withdraw from the study at any time.
* What treatments or interventions did the participants take/receive? Participants were randomly assigned to one of four study groups: P4M3 CA35, P4M3 CM35, Cigarette, or smoking abstinence, for five days in a confinement setting. Participants assigned to one of the P4M3 arms or the Cigarette arm could use their assigned product at will and as often as they desired during the five-day confinement period. Participants assigned to the smoking abstinence arm had to abstain from cigarette smoking. Urine was collected from each participant for harmful and potentially harmful constituent analysis, for each 24 hours, from Day 1 (i.e., the start of the confinement period) to Day 5 (until discharge at the morning of Day 6). Participants were also asked to evaluate their experience of using their assigned products, using the Product Evaluation Scale (PES) questionnaire. The PES assessed the degree to which subjects experienced the 'reinforcing effects' of the use of P4M3 for both flavour variants in cigarette smokers switching to P4M3 compared to subjects continuing cigarette smoking. The PES is composed of five scales which address the degree to which participants experienced different effects (Product Satisfaction, Psychological Rewards, Aversion, Enjoyment of respiratory tract sensations, and Craving Reduction) as a result of using the P4M3 or the cigarette, rated on a 7 point scale from 1 = "not at all" to 7 = "extremely."
* What medical problems (adverse reactions) did the participants have? Overall, during the product use, 23 adverse reactions occurred in 17 participants, all of them being mild or moderate in severity. Only one adverse reaction (oropharyngeal pain) was considered related to an investigational product (P4M3 CM35) and occurred in just one participant. There were no clinically significant findings in the physical examination, clinical laboratory, vital signs, or ECG assessments in this study.
* What happened during the study? A presentation of P4M3 (without product use) was made to the participants during the Screening visit. All participants received information on the risks of smoking, smoking cessation advice, and a briefing that the use of P4M3 is not risk-free. Eligible participants, fulfilling all criteria for participation, returned to the investigational site for confirmation of eligibility at the Admission visit (Day -2). On Day -2 (Admission), after eligibility criteria had been verified, all eligible participants were enrolled and performed a product test using both P4M3 flavour variants for a duration of approximately 10 minutes use per variant. After the product test, subjects not willing to use P4M3 during the study were to be discontinued and be replaced. Participants willing to continue their participation in the study started their confinement period. On Day -1, participants were randomly assigned to one of four arms: P4M3 CA35 variant; P4M3 CM35 variant; Cigarettes; Smoking Abstinence. Participants were informed about their randomization arm by the study site staff on Day 1 prior to the start of product use. The Exposure period in confinement began on Day 1 and consisted of 5 days of at will use of the assigned product in the P4M3 and Cigarette arms. Use of any tobacco/nicotine containing product other than the assigned product was not allowed and, at the discretion of the study doctor, resulted in the participant's discontinuation from the study. Participants allocated to the Smoking Abstinence arm had to abstain from Cigarette smoking. Daily 24-hour urine was collected from Day 1 to Day 5 for harmful and potentially harmful constituent analysis. On Day 1, use of P4M3 or Cigarette smoking in the respective arms was not supposed to start before the end of 24-hour urine collection of Day -1. The 24 hour urine collection period for Day 5 ended in the morning of Day 6 prior to Discharge. On Day -1 and on Days 1 to 5, participants completed questionnaires about product evaluation, craving, and liking assessments. During the confinement period, site staff distributed assigned products to the participants and recorded all distributed products in the participants' files. Any participant who wanted to attempt to quit using any tobacco or nicotine-containing product at any time during the study (that is, to quit P4M3 use or Cigarette smoking) was encouraged to do so and was to be referred to appropriate medical services. This decision would not affect the participant's financial compensation, and the participant was to be considered as remaining in the study. The Exposure period to the assigned investigational product (P4M3 or Cigarette) ended at 11:00 PM on Day 5, followed by Discharge on Day 6 after completion of all study procedures. Participants were allowed to smoke Cigarettes or use other tobacco or nicotine-containing products, at their discretion, only after discharge from the study. After discharge at Day 6 or from the day of an early termination, subjects entered a 3-day Safety follow-up period during which any adverse reactions reported by the participants were collected. The follow-up of adverse reactions ongoing at discharge was conducted by the investigational site.
* What were the results of the study? The results of this study demonstrated that switching exclusively from cigarettes to the P4M3 electronic nicotine delivery system for five days resulted in substantial reductions in exposure to the harmful and potentially harmful constituents of cigarette smoke, while maintaining comparable levels of nicotine exposure. The harmful and potentially harmful constituents of cigarette smoke were examined by measuring their degradation products in participant's urine. These degradation products are called Biomarkers of Exposure. As another Biomarker of Exposure, the saturation of hemoglobin in the blood with carbon monoxide was measured. The magnitude of reduction in the levels of Biomarkers of Exposure were comparable between both variants of P4M3 (CA35 tobacco flavour and CM35 menthol flavour). The reductions observed for most of the Biomarker of Exposure levels in the P4M3 arms, in timing as well as in magnitude, approached those levels observed for smoking abstinence. Furthermore, no additional safety concerns were associated with P4M3 compared to cigarette smoking or smoking abstinence.
* How has this study helped patients and researchers? The participants in this study were healthy, current cigarette smokers. All participants were informed about the health risks associated with smoking and were given smoking cessation advice. Participants in this clinical study benefited from repeated and detailed general health check-ups. This clinical study may help doctors and scientists learn about electronic nicotine delivery systems. The exposure period in confinement provided information on the exposure reductions achievable for harmful and potentially harmful constituents in a well-controlled environment with full control over daily P4M3 and/or Cigarette consumption, compared to smoking abstinence.
* Details of any further research planned: There is currently no further research planned with P4M3 Generation 2.0.

ELIGIBILITY:
Main Inclusion Criteria:

* Subject has signed the Informed Consent Form (ICF) and is able to understand the information provided in the ICF.
* Subject has been a smoker for ≥3 years prior to the screening visit (smoking cessation attempts during this period, if any, did not last >6 months).
* Subject has continuously smoked on average ≥10 commercially available mentholated or non-mentholated CIGs per day over the last 4 weeks prior to screening and admission. Smoking status will be verified based on a urinary cotinine test (cotinine ≥200 ng/mL).
* Subject is healthy as judged by the Investigator based on available assessments from the screening period (e.g., safety laboratory, spirometry, vital signs, physical examination, ECG, and medical history).

Main Exclusion Criteria:

* Subject has a clinically relevant disease which requires medication (including but not limited to gastrointestinal, renal, hepatic, neurological, hematological, endocrine, oncological, urological, immunological, pulmonary, and cardiovascular disease) or any other medical condition (including safety laboratory), which as per the judgment of the Investigator would jeopardize the safety of the subject.
* Subject experienced within 30 days prior to screening/admission a body temperature >37.5°C or an acute illness (e.g., upper respiratory-tract infection, viral infection, etc.)
* As per the Investigator's judgment, the subject has medical conditions which do or will require a medical intervention (e.g., start of treatment, surgery, hospitalization) during the study participation, which may interfere with the study participation and/or study results.
* Subject has relevant history of a current asthma condition or chronic obstructive pulmonary disease (COPD) condition, and/or clinically significant spirometry findings at Screening or Baseline
* Subject has donated blood or received whole blood or blood products within 3 months prior to screening.
* BMI <18.5 kg/m2 or ≥32.0 kg/m2.

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2022-07-15 (Actual); Primary Completion 2022-08-31 (Actual); Study Completion 2022-11-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Patrick Winiger, MD, Principal Investigator — Celerion
Locations (1):
- Celerion, Belfast, United Kingdom

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | P4M3 CA35 | P4M3 CM35 | Cigarette | Smoking Abstinence
Started | 16 | 17 | 18 | 17
Completed | 16 | 17 | 17 | 17
Not Completed | 0 | 0 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Enrolled But Not Randomized: Subjects enrolled in the study but not randomized.
- Total: Total of all reporting groups
Arm/Group | P4M3 CA35 | P4M3 CM35 | Cigarette | Smoking Abstinence | Enrolled But Not Randomized | Total
Number analyzed (Participants) | 16 | 17 | 18 | 17 | 6 | 74
Age, Continuous [Mean (Standard Deviation); unit: years] | 39.5 (11.69) | 40.3 (11.49) | 39.8 (11.75) | 38.6 (10.03) | 39.7 (10.07) | 39.6 (10.89)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 8 | 8 | 8 | 0 | 31
  Male | 9 | 9 | 10 | 9 | 6 | 43
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 1 | 0 | 0 | 0 | 0 | 1
  White | 15 | 17 | 18 | 17 | 6 | 73
  More than one race | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
BMI at admission [Mean (Standard Deviation); unit: kg/m²] | 25.46 (2.316) | 25.74 (3.486) | 24.98 (2.963) | 24.54 (2.769) | 26.12 (1.513) | 25.25 (2.812)

OUTCOME MEASURES:

1. Primary Outcome: 3-HPMA
Description: To measure change in 3-hydroxypropyl mercapturic acid (3-HPMA), which is a biomarker of exposure to Acrolein.
Time Frame: From baseline to 5 days
Population: Some participants were excluded from analysis for protocol deviations (including, but not limited to, missing measurements).
Measure: Geometric Mean (95% Confidence Interval); unit: ng/mg creatinine
Arm/Group | P4M3 CA35 | P4M3 CM35 | Cigarette | Smoking Abstinence
Number analyzed (Participants) | 16 | 16 | 18 | 16
ng/mg creatinine
  Baseline | 657.46 [469.82 to 920.03] | 726.84 [536.06 to 985.51] | 703.29 [544.68 to 908.10] | 724.06 [516.52 to 1015.00]
  After 1 day of exposure | 154.27 [120.24 to 197.92] | 155.85 [131.79 to 184.30] | 638.77 [486.69 to 838.37] | 149.66 [121.66 to 184.11]
  After 2 days of exposure: number analyzed (Participants) | 16 | 16 | 18 | 15
  After 2 days of exposure | 171.00 [144.04 to 203.00] | 167.93 [141.24 to 199.66] | 794.49 [621.70 to 1015.29] | 147.57 [119.15 to 182.76]
  After 3 days of exposure | 112.48 [91.31 to 138.56] | 109.29 [97.88 to 122.02] | 670.16 [496.06 to 905.36] | 93.16 [82.69 to 104.96]
  After 4 days of exposure: number analyzed (Participants) | 16 | 15 | 18 | 16
  After 4 days of exposure | 194.46 [155.93 to 242.50] | 241.24 [189.75 to 306.70] | 728.51 [549.25 to 966.27] | 189.48 [154.44 to 232.46]
  After 5 days of exposure: number analyzed (Participants) | 15 | 16 | 17 | 16
  After 5 days of exposure | 105.20 [90.85 to 121.83] | 111.12 [89.54 to 137.90] | 544.77 [373.74 to 794.07] | 93.20 [81.69 to 106.34]

2. Primary Outcome: 2-CyEMA
Description: To measure change in 2-cyanoethyl mercapturic acid (2-CyEMA), which is a biomarker of exposure to Acrylonitrile.
Time Frame: From baseline to 5 days
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: ng/mg creatinine
Arm/Group | P4M3 CA35 | P4M3 CM35 | Cigarette | Smoking Abstinence
Number analyzed (Participants) | 16 | 16 | 18 | 16
ng/mg creatinine
  Baseline | 97.17 [69.12 to 136.61] | 108.50 [81.79 to 143.92] | 98.85 [77.25 to 126.50] | 100.39 [70.02 to 143.92]
  After 1 day of exposure | 33.47 [22.35 to 50.12] | 37.47 [28.39 to 49.44] | 90.13 [69.22 to 117.34] | 33.68 [22.17 to 51.18]
  After 2 days of exposure: number analyzed (Participants) | 16 | 16 | 18 | 15
  After 2 days of exposure | 17.99 [10.93 to 29.60] | 22.95 [17.71 to 29.75] | 100.04 [77.18 to 129.66] | 18.12 [10.05 to 32.66]
  After 3 days of exposure | 16.40 [9.08 to 29.61] | 20.06 [14.91 to 26.98] | 96.41 [71.29 to 130.38] | 15.67 [8.52 to 28.82]
  After 4 days of exposure: number analyzed (Participants) | 16 | 15 | 18 | 16
  After 4 days of exposure | 12.79 [7.26 to 22.55] | 16.78 [12.70 to 22.19] | 85.54 [61.48 to 119.02] | 14.40 [8.08 to 25.64]
  After 5 days of exposure: number analyzed (Participants) | 15 | 16 | 17 | 16
  After 5 days of exposure | 12.31 [6.81 to 22.25] | 17.09 [11.93 to 24.47] | 79.87 [54.04 to 118.05] | 12.95 [7.02 to 23.87]

3. Primary Outcome: Total NNAL
Description: To measure change in Total 4-(methylnitrosamino)-1-(3-pyridyl)-1-butanol (total NNAL), which is a biomarker of exposure to 4-(methylnitrosamino)-1-(3- pyridyl)-1-butanone (NNK).
Time Frame: From baseline to 5 days
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: pg/mg creatinine
Arm/Group | P4M3 CA35 | P4M3 CM35 | Cigarette | Smoking Abstinence
Number analyzed (Participants) | 16 | 16 | 18 | 16
pg/mg creatinine
  Baseline | 114.66 [71.39 to 184.15] | 145.13 [96.82 to 217.53] | 116.41 [78.30 to 173.06] | 115.95 [66.28 to 202.86]
  After 1 day of exposure | 58.27 [32.64 to 104.03] | 85.16 [58.39 to 124.22] | 106.12 [69.17 to 162.81] | 68.39 [39.47 to 118.50]
  After 2 days of exposure: number analyzed (Participants) | 16 | 16 | 18 | 15
  After 2 days of exposure | 46.46 [26.01 to 82.96] | 63.61 [40.95 to 98.82] | 112.97 [75.73 to 168.53] | 44.14 [20.37 to 95.65]
  After 3 days of exposure | 42.80 [22.50 to 81.41] | 59.25 [36.83 to 95.32] | 111.82 [74.08 to 168.79] | 40.39 [20.14 to 80.99]
  After 4 days of exposure: number analyzed (Participants) | 16 | 15 | 18 | 16
  After 4 days of exposure | 36.24 [19.60 to 66.99] | 51.10 [32.64 to 80.02] | 102.41 [66.16 to 158.52] | 37.82 [18.68 to 76.57]
  After 5 days of exposure: number analyzed (Participants) | 15 | 16 | 17 | 16
  After 5 days of exposure | 32.73 [17.63 to 60.78] | 53.87 [32.16 to 90.23] | 101.05 [64.72 to 157.78] | 37.94 [18.91 to 76.12]

4. Primary Outcome: COHb
Description: To measure change in carboxyhemoglobin (COHb), which is a biomarker of exposure to Carbon monoxide (CO).
Time Frame: From baseline to 5 days
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: percent saturation of hemoglobin
Arm/Group | P4M3 CA35 | P4M3 CM35 | Cigarette | Smoking Abstinence
Number analyzed (Participants) | 16 | 16 | 18 | 16
percent saturation of hemoglobin
  Baseline | 2.99 [2.53 to 3.53] | 2.91 [2.38 to 3.54] | 2.58 [2.36 to 2.83] | 2.71 [2.40 to 3.07]
  After 1 day of exposure: number analyzed (Participants) | 16 | 15 | 18 | 16
  After 1 day of exposure | 3.06 [2.60 to 3.60] | 3.10 [2.45 to 3.92] | 2.69 [2.47 to 2.93] | 2.96 [2.56 to 3.43]
  After 2 days of exposure: number analyzed (Participants) | 16 | 16 | 18 | 15
  After 2 days of exposure | 1.71 [1.58 to 1.86] | 1.80 [1.52 to 2.13] | 2.87 [2.64 to 3.12] | 1.64 [1.55 to 1.75]
  After 3 days of exposure: number analyzed (Participants) | 16 | 16 | 18 | 15
  After 3 days of exposure | 1.55 [1.43 to 1.68] | 1.59 [1.48 to 1.71] | 2.80 [2.53 to 3.10] | 1.57 [1.44 to 1.71]
  After 4 days of exposure | 1.64 [1.39 to 1.95] | 1.69 [1.38 to 2.07] | 2.72 [2.44 to 3.03] | 1.45 [1.33 to 1.57]
  After 5 days of exposure: number analyzed (Participants) | 16 | 16 | 17 | 16
  After 5 days of exposure | 1.52 [1.41 to 1.63] | 1.53 [1.39 to 1.68] | 2.78 [2.45 to 3.15] | 1.45 [1.26 to 1.67]

ADVERSE EVENTS:
Time Frame: Adverse events were collected from the signature of the ICF by each subject until the end of the safety follow-up period, a total duration for each subject of up to 38 days.
Arm/Group | P4M3 CA35 | P4M3 CM35 | Cigarette | Smoking Abstinence | Enrolled But Not Randomized
All-Cause Mortality (participants affected / at risk) | 0/16 | 0/17 | 0/18 | 0/17 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/17 | 0/18 | 0/17 | 0/6
Other Adverse Events (participants affected / at risk) | 1/16 | 5/17 | 4/18 | 6/17 | 1/6
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | P4M3 CA35 (N=16) | P4M3 CM35 (N=17) | Cigarette (N=18) | Smoking Abstinence (N=17) | Enrolled But Not Randomized (N=6)
Headache (Nervous system disorders) | 0 (0) | 1 (1) | 3 (3) | 2 (2) | 1 (1)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Arthropod Sting (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Skin laceration (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pain (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dysmenorrhoea (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
We confirm we have the contractual provisions in place which specify that in no event will the study site be allowed to disclose to any third party (or publicly release) any information obtained through the study without the CRO's prior written consent which in turn cannot provide such consent without Sponsor's approval unless such publication is made to satisfy regulatory requirements.

The Intellectual Property rights and research results from the present study belong to the Sponsor.

DOCUMENTS (2):
  • Study Protocol (2022-04-13): https://cdn.clinicaltrials.gov/large-docs/56/NCT05487456/Prot_000.pdf
  • Statistical Analysis Plan (2022-08-26): https://cdn.clinicaltrials.gov/large-docs/56/NCT05487456/SAP_001.pdf